CLINICAL TRIAL: NCT06506890
Title: C-POLAR System Intervention in a Long-Term Care Facility HVAC Filter Study (C-Polar LTC)
Brief Title: Study to Determine the Difference in Reduction of Bioaerosols in a Long-term Care Facility
Acronym: C-PolarLTC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C-Polar Innovations (Industry)
Collaborators: Kelowna General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H23-04137
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Air Pollution
Keywords: Long-term care; Air Quality; HVAC Filter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- comparing the difference in reduction of bioaerosols between HVAC filters (Other): comparing the difference in reduction of bioaerosols between HVAC filters.
  Interventions: Other: Use of C-Polar coated HVAC Filter versus conventional HVAC Filter

INTERVENTIONS:
Other: Use of C-Polar coated HVAC Filter versus conventional HVAC Filter — comparing the difference in reduction of bioaerosols between HVAC filters.
  Other Names: comparing the difference in reduction of bioaerosols between HVAC filters.

SUMMARY:
This is a CONTROLLED PROSPECTIVE COHORT study of a long-term care facility. At the start of the study a dedicated section A of the facility ventilation system will have routine HVAC filters of the same dimensions installed, while section B of the same facility ventilation system will have C-POLAR (cationic polymeric coated) HVAC filters installed. There will be continuous Indoor Air Quality monitors (PM 2.5, CO2, VOC, Radon, Temp, and RH) installed at different vent locations throughout the long-term care facility for the duration of the study. Air samples with an Airport MD8 BAMS machine will be taken once a week at various vent locations at the long-term care facility.

DETAILED DESCRIPTION:
This is a CONTROLLED PROSPECTIVE COHORT study of a long-term care facility. At the start of the study a dedicated section A of the facility ventilation system will have routine HVAC filters of the same dimensions installed, while section B of the same facility ventilation system will have C-POLAR (cationic polymeric coated) HVAC filters installed. There will be continuous Indoor Air Quality monitors (PM 2.5, CO2, VOC, Radon, Temp, and RH) installed at different vent locations throughout Cottonwoods for the duration of the study. Air samples with an Airport MD8 BAMS machine will be taken once a week at various vent locations at the long-term care facility. The aim of this study is to determine the difference in reduction of bioaerosols in a long-term care facility with MERV 13 C-POLAR (cationic polymeric coated) HVAC filters compared to conventional MERV 13 HVAC filters.

Primary Endpoint:

This study aims to determine the reduction of bioaerosols (BAMS) in a facility with a C-POLAR HVAC filter building intervention versus conventional filters.

Secondary Endpoints:

1. Volatile organic compound (VOC)
2. Radon determination
3. Static, passive particulate determination from air
4. Air microbiome analysis
5. Air Quality and Respiratory Staff Survey

Radon gas testing, particulate matter testing (PM2.5) [fine inhalable particles, with diameters that are generally 2.5 micrometers and smaller]. Carbon dioxide testing (CO2), VOCs testing [volatile organic compounds (airborne chemicals)], relative humidity (RH) testing [it is a measure of the actual amount of water vapor in the air compared to the total amount of vapor that can exist in the air at its current temperature], and temperature readings.

ELIGIBILITY:
Inclusion Criteria:

1. Any resident, staff, and any individual who enters the long term care facility will be in a broad sense, involved in this study, as the MERV 13 HVAC filters will be installed within the HVAC system and will not allow anyone to not participate in the study who enters the facility. It is impracticable to carry out this research of comparing two different HVAC filters in an active long term care setting by receiving prior consent from all individuals who may enter, such as vendors or visitors. This research involves no more than minimal risk and may or may not improve air quality or minimize bioaerosols in the facility.

Exclusion Criteria:

1. Does not wish to enter the long-term care facility until completion of study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is comparing the difference in reduction of bioaerosols between MERV 13 HVAC filters. | Nine Months
  The aim of this study is to determine the difference in reduction of bioaerosols in a long-term care facility with MERV 13 C-POLAR (cationic polymeric coated) HVAC filters compared to conventional MERV 13 HVAC filters.

CONTACTS AND LOCATIONS:
Overall Officials: Deanne Taylor, PhD, Principal Investigator — Kelowna General Hospital; Michael Mansour, MD, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Kelowna General Hospital, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
All participant data will be anonymized